CLINICAL TRIAL: NCT05825482
Title: Breast Margin Study: Routine Cavity Shave Margins Vs. Selective Margins Using Savi Scout®
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE5122
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Savi Scout; Shave margin; Selective margin; Breast-Q
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Partial mastectomy with Savi Scout® localization and routine cavity shave margins
  Interventions: Procedure: Arm 1 Partial mastectomy with Savi Scout® localization and shave margins.
- Arm 2 (Active Comparator): Partial mastectomy with Savi Scout® localization and selective shave margins.
  Interventions: Procedure: Arm 2 Partial mastectomy with Savi Scout® localization and selective shave margins.

INTERVENTIONS:
Procedure: Arm 1 Partial mastectomy with Savi Scout® localization and shave margins. — Patients will undergo preoperative Savi Scout® reflector placement under image guidance per routine care. Patients will undergo randomization. With Arm 1 randomization, the surgeons will be instructed to perform a partial mastectomy with routine cavity shave margins using Savi Scout® localization. The lesion will be removed in the routine fashion. The surgeons will use the Savi Scout® to perform routine cavity shave margins by extracting superior, lateral, inferior, medial, anterior, and posterior margins.
  Arms: Arm 1
Procedure: Arm 2 Partial mastectomy with Savi Scout® localization and selective shave margins. — Patients will undergo preoperative Savi Scout® reflector placement under image guidance per routine care. Patients will undergo randomization. With Arm 2 randomization, the surgeons will be instructed to perform a partial mastectomy with selective margins shave margins using Savi Scout®. The lesion will be removed in the routine fashion. The Savi Scout® localizer will be utilized to determine selective shave margins by examining the same margins on the excised tissue specimen. The surgeon will obtain selective margins if the margin of the tissue specimen is within 1mm of invasive cancer and 2mm within DCIS.
  Arms: Arm 2

SUMMARY:
This is a prospective study comparing partial mastectomy performed with routine cavity shave margins and Savi Scout® localization to partial mastectomy performed with selective margins and Savi Scout® localization. The primary objective is to determine the difference in positive margin rate between the two methods. The secondary objectives are to determine the differences in the rate of re-excision, volume of tissue extracted and Breast-Q® score between the two methods. It is hypothesized that the Savi Scout® will allow for decreased volume of tissue excised when compared to routine cavity shave margins without any difference in positive margin rate or rate of re-excision.

DETAILED DESCRIPTION:
Over a period of 24 months, this study will recruit 204 women 18 years and older with stage I-II breast cancer or stage 0 DCIS that have been diagnosed by core needle biopsy and are planning to receive breast conserving surgery.

After obtaining consent, the patient will be asked to complete the Breast-Q® questionnaire which should take about 10-15 minutes for the patient to complete. The patient will then be randomized in a 1:1 fashion to:

Arm 1: Partial mastectomy with Savi Scout® localization and routine cavity shave margins

Arm 2: Partial mastectomy with Savi Scout® localization and selective shave margins.

Arm 1 and 2 patients will undergo preoperative Savi Scout® reflector placement under image guidance per routine care. The surgeons will be instructed to perform a partial mastectomy with routine cavity shave margins using Savi Scout® or partial mastectomy with selective margins using Savi Scout®. The lesion will be removed in the routine fashion. For patients in arm 1, the surgeons will use the Savi Scout® to perform routine cavity shave margins by extracting superior, lateral, inferior, medial, anterior, and posterior margins. For patients in arm 2, the Savi Scout® localizer will be utilized to determine selective shave margins by examining the same margins on the excised tissue specimen. The surgeon will obtain selective margins if the margin of the tissue specimen is within 1mm of invasive cancer and 2mm within DCIS. All surgeons participating in the study will undergo an educational session to ensure consistency.

Tissue specimens will be processed per hospital policy and sectioned for gross evaluation. Tissue specimens will be assessed by the pathologists at Cleveland Clinic Akron General. This simulates typical pathology review. Positive margin rate is a categorical variable and will be reviewed by pathology board certified physicians and thus should have minimal interpersonal variation.

At the postoperative visit, the patient will be asked to complete another Breast-Q® questionnaire.

ELIGIBILITY:
Inclusion Criteria

* Women 18 years and older, and
* With Clinical stage I-II invasive breast cancer, or Stage 0 DCIS, and
* That have been diagnosed by means of core needle biopsy appropriate for breast conserving therapy, and
* Present to Cleveland Clinic Akron General.
* Subjects must have pathologically confirmed breast carcinoma or ductal carcinoma in situ.
* Performance status: ECOG 0-1
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Patients may have received or may be receiving endocrine therapy.

Exclusion Criteria

* Men
* Pregnant women
* Patients who have received neoadjuvant chemotherapy for current cancer diagnosis.
* Patients with current diagnosis of synchronous bilateral breast cancer. (A diagnosis of breast cancer at least one year prior to current cancer diagnosis is acceptable.)
* Patients < 18 years of age.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 204 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Determine the difference in positive margin rate between the two methods. | 24 months
  The primary objective is to determine the difference in positive margin rate between the two methods.

SECONDARY OUTCOMES:
Difference in the rate of re-excision between the two methods. | 24 months
  Determine the difference in the rate of re-excision between the two methods.
Difference in the volume of tissue extracted between the two methods. | 24 months
  Determine the difference in the volume of tissue extracted between the two methods.
Difference in the BREAST-Q® Version 2.0 Breast Conserving Therapy Module Pre- and Postoperative Scales | 24 months
  Determine the difference in the Breast-Q® scores between the two methods. Scores range from 0 (worst) to 100 (best). Higher scores reflect a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Fenton, M.D., Principal Investigator — Cleveland Clinic Akron General, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Akron General, Case Comprehensive Cancer Center, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No